CLINICAL TRIAL: NCT06633003
Title: Effects of Oral Administration of Antrodia Cinnamomea Products for Clinical Symptoms in Spinocerebellar Ataxia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ALPS Biotech CO. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 202404011RSA
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Spinocerebellar Ataxia
Keywords: Neuroinflammatory Diseases; Nervous System Diseases; Spinocerebellar Ataxia; Antrodia Cinnamomea
MeSH Terms: conditions — Spinocerebellar Ataxias; Neuroinflammatory Diseases; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Placebo-controlled crossover design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage I: Antrodia Cinnamomea Products + Stage II: Placebo (Active Comparator): Crossover design:
  During 0 week~8 weeks is Stage I :
  • Dietary Supplement: Antrodia Cinnamomea Products
  During 16 weeks~ 24 weeks is Stage II:
  • Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Antrodia cinnamomea Products
- Stage I: Placebo + Stage II: Antrodia Cinnamomea Products (Placebo Comparator): Crossover design:
  During 0 week~8 weeks is Stage I :
  • Dietary Supplement: Placebo
  During 16 weeks~ 24 weeks is Stage II:
  • Dietary Supplement: Antrodia Cinnamomea Products
  Interventions: Dietary Supplement: Antrodia cinnamomea Products

INTERVENTIONS:
Dietary Supplement: Antrodia cinnamomea Products — Placebo-controlled crossover design:
  * Dietary Supplement: Antrodia Cinnamomea Products
  * Dietary Supplement: Placebo
  Arms: Stage I: Antrodia Cinnamomea Products + Stage II: Placebo
Dietary Supplement: Antrodia cinnamomea Products — A arm :
  Stage I :
  • Dietary Supplement: Antrodia Cinnamomea Products
  Stage II:
  • Dietary Supplement: Placebo
  B arm :
  Stage I :
  • Dietary Supplement: Placebo
  Stage II:
  • Dietary Supplement: Antrodia Cinnamomea Products
  Arms: Stage I: Placebo + Stage II: Antrodia Cinnamomea Products

SUMMARY:
This study aims to assess the effect of Antrodia cinnamomea on clinical symptoms in spinocerebellar ataxia patients. To investigate the advancements in neurodegenerative diseases.

DETAILED DESCRIPTION:
This study aims to assess the effect of Antrodia cinnamomea on clinical symptoms in spinocerebellar ataxia patients: a randomized, double-blind, placebo-controlled crossover design, and parallel clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 30 to 70 years, whose native language is Chinese.
2. Patients diagnosed with Spinocerebellar Ataxia.
3. Subjects with a score below 30 on the Scale for the Assessment and Rating of Ataxia (SARA scale).
4. Individuals who can read and write in Chinese and communicate in Chinese.
5. Agree to participate in the study.

Exclusion Criteria:

1. Patients with severe systemic diseases, such as heart or respiratory failure, liver or kidney failure, severe brain injury, prolonged bed rest, or incurable malignancies.
2. Pregnant women and breastfeeding mothers.
3. Patients who have taken Antrodia cinnamomea products within the last 6 months prior to the trial.
4. Patients with other factors that prevent them from continuing to participate in this study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the total score of the Scale for the Assessment and Rating of Ataxia (SARA) at 48 weeks in subjects is compared to natural history. | Up to 48 weeks of treatment.
  To compare the effectiveness of Antrodia Cinnamomea Products in treating SCA, as measure by the Scale for the Assessment and Rating of Ataxia (SARA), in subjects randomized to treatment after 24 weeks of treatment. The SARA is a scale with a range of 0 to 40, where an increase in the total score indicates a worsening of symptoms.

SECONDARY OUTCOMES:
Resting-state electroencephalogram (EEG) will be collected | Up to 48 weeks of treatment.
  Successful attainment of Resting-state electroencephalogram (EEG). To compare the EEG recordings in different frequency band change before, during, and after the Antrodia Cinnamomea Products used.
Collect Cytokines assay of plasma exosomes and Neurofilament Light Chain (NfL) Test of plasma. | Up to 48 weeks of treatment.
  Monitor Cytokines assay of plasma exosomes and Neurofilament Light Chain (NfL) Test of plasma.
The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses. | Up to 48 weeks of treatment.
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses.
  The evaluator should start the stopwatch as soon as the patient touches the first peg. The evaluator should stop the stopwatch once the last peg is in the container.
  Scoring:
  The number of seconds it takes for the patient to complete the test, where an increase in the total score indicates a worsening of symptoms.
Changes From Start of Administration (Week 0) in Pittsburgh Sleep Quality Index (PSQI) Global Score at End of Study. | Up to 48 weeks of treatment.
  PSQI is a self-rated questionnaire for sleep quality. It includes 18 items across 7 components; C1: Sleep quality, C2: Sleep latency, C3: Sleep duration, C4: Sleep efficiency, C5: Sleep disturbance, C6: Use of sleep medication, C7: Daytime dysfunction. Each component is scored 0-3 (0 = no difficulty, 3=severe difficulty), and total score ranging from 0 to 21. It included seven components with a global PSQI score > 5 is indicative of poor sleep quality.
Hospital Anxiety and Depression Scale (HADS) | Up to 48 weeks of treatment.
  Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
The 8 Metre Walk Test. | Up to 48 weeks of treatment.
  The 8 Metre Walk Test is a performance measure used to assess walking or gait speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function
  Scoring The total time taken to ambulate 8 meters is recorded. Timing starts when the toes pass the 0-meter mark. Timing stops when the toes pass the 8-meter mark. The 8-meter is then divided by the total time taken (in seconds) to completed. Increase in the total time indicates a worsening of symptoms.

OTHER OUTCOMES:
Check Fecal levels of Human Calprotectin and Fecal levels of Human Lactoferrin. | Up to 48 weeks of treatment.
  Check Fecal levels of Human Calprotectin and Fecal levels of Human Lactoferrin.

CONTACTS AND LOCATIONS:
Overall Officials: MingChe Kuo, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No